## **Informed Consent Form**

Official Title: Combined Muscle Energy
Technique and Myofascial Chain
Stabilization Reduces Menstrual Pain and
Improves Pelvic Alignment in Women With
Primary Dysmenorrhea: A Prospective Study

**NCT Number: [Pending]** 

Date: December 10, 2024

Informed Consent Form

Combined Muscle Energy Technique and Myofascial Chain Stabilization Reduces

Menstrual Pain and Improves Pelvic Alignment in Women With Primary

Dysmenorrhea: A Prospective Study

NCT Number: [Pending]

Document Date: December 10, 2024

1. Introduction

You are invited to participate in a research study evaluating the effects of Muscle

Energy Technique (MET) combined with myofascial chain-based pelvic stabilization

training on pelvic alignment and menstrual pain in women diagnosed with primary

dysmenorrhea. This document provides information to help you decide whether or

not to participate.

2. Purpose of the Study

The purpose of this study is to determine whether MET combined with pelvic

stabilization training can reduce pain and improve pelvic alignment in women with

moderate to severe primary dysmenorrhea.

3. Procedures

If you agree to participate, you will be assigned to either the experimental group

(receiving a combination of Muscle Energy Technique [MET] for iliac and sacral

dysfunctions [20 minutes] and myofascial chain-based pelvic stabilization training

[30 minutes]), or the control group (receiving medium- and low-frequency

interferential current therapy [ICT, 20 minutes] and deep friction massage [DFM, 30

minutes] targeting the lumbar, sacroiliac, and iliac crest regions). Each session will

last 50 minutes, delivered 3 times per week for 4 weeks. Assessments will be

conducted at baseline, after 4 weeks, and at a 12-week follow-up via telephone.

4. Risks and Discomforts

There are minimal risks associated with this study. You may experience temporary

muscle soreness or fatigue following treatment sessions. All procedures will be

conducted by trained professionals.

5. Benefits

Potential benefits include relief from menstrual pain, improved posture, and better

pelvic alignment. However, these outcomes are not guaranteed.

6. Confidentiality

All personal and medical information will be kept confidential. Your identity will not

be revealed in any publication or presentation resulting from this study.

7. Voluntary Participation

Participation in this study is voluntary. You may refuse to participate or withdraw at

any time without penalty or loss of benefits.

8. Contact Information

If you have questions about the study, please contact:

Shanjiao Luo (Principal Investigator)

Email: luoshanjiao@gmail.com

Affiliation: Department of Rehabilitation, Shenzhen JianAn Hospital

9. Consent

By signing below, you agree that you have read and understood this document and

voluntarily consent to participate in the study.

| Participant Name: _ | |
|---------------------|---|
| - | |
| Signature: | |
| | • |
| Date: | |